CLINICAL TRIAL: NCT01113372
Title: Optimized Duration of Clopidogrel Therapy Following Treatment With the Endeavor Zotarolimus - Eluting Stent in the Real World Clinical Practice - Optimize Trial
Brief Title: Optimized Duration of Clopidogrel Therapy Following Treatment With the Endeavor - Optimize Trial
Acronym: OPTIMIZE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cardiovascular Research Center, Brazil (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OPTIMIZE
Record Dates: First submitted 2010-04-22; First posted 2010-04-29 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary, Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel 3 months (Experimental): Regime of dual antiplatelet therapy (DAPT) including aspirin+clopidogrel for 3 months.
  Interventions: Drug: Clopidogrel
- Clopidogrel 12 months (Active Comparator): Regime of dual antiplatelet therapy (DAPT) including aspirin+clopidogrel for 12 months.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 75mg daily.

SUMMARY:
Prospective, multicenter, randomized (two-arm 1:1), non-inferiority clinical evaluation comparing 2 regimes of dual antiplatelet therapy (DAPT) with aspirin + clopidogrel following percutaneous coronary intervention (PCI) with Endeavor Zotarolimus eluting stent (ZES) to evaluate the impact of different regimes of DAPT on clinical outcomes in minimally selected patients from the "real-world" clinical practice receiving the Endeavor ZES for the treatment of coronary artery lesions. Patients undergoing percutaneous treatment with the Endeavor ZES will be randomized in a 1:1 ratio to 2 regimens of DAPT including oral clopidogrel 75mg/day for 3 months versus 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. patients >18 years of age,
2. clinical indication for PCI with stent implantation of at least one angiographically documented coronary artery lesion,
3. agreement to undergo all protocol clinical follow-ups. 4 - presence of at least one obstruction >50% diameter stenosis by visual estimation in a major epicardial vessel or a major branch (≥2.50mm), with coronary anatomy suitable for percutaneous treatment with implantation of the Endeavor ZES.

Exclusion Criteria:

1. ST-elevation acute MI presenting for primary or rescue PCI;
2. DES in-stent restenosis;
3. PCI with bare metal stents <6 months prior to index procedure;
4. previous treatment with any DES;
5. scheduled elective surgery within 12 months post index procedure;
6. contra-indication, intolerance, or known hypersensibility to aspirin and/or clopidogrel;
7. known illness with life expectancy <36 months; and impossibility to comply with all protocol follow-ups.
8. target lesion(s) located in saphenous vein grafts,
9. coronary anatomy unsuitable for percutaneous treatment with implantation of the Endeavor ZES.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3119 (Actual)
Dates: Start 2010-04; Primary Completion 2013-02 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
NACCE | 12 months clinical follow-up
  rates of Net Clinical Benefit (net adverse clinical and cerebral events, NACCE) at 12 months clinical follow-up. The primary endpoint is defined as the composite endpoint of: death by any cause, myocardial infarction (MI), cerebral vascular accident, and major bleeding (according to the modified REPLACE-2 and GUSTO criteria). The primary endpoint will be assessed only in patients receiving exclusively the Endeavor ZES during index (and staged) procedure.

SECONDARY OUTCOMES:
Rates of Stent thrombosis | until 24 and 36 months
Target vessel revascularization (TVR) and target lesion revascularization (TLR) | 6 and 12 months
MACE (major adverse cardiac events) at in-hospital, 30 days, 6, 12, 18, 24 and 36 months; DAPT compliance (according to treatment allocation in the trial) | until 36 months
Major bleeding according to the modified REPLACE-2 and GUSTO criteria events at 1, 3, 6 and 12 months follow-up | until 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Feres, PhD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia
Locations (32):
- Brazil (32):
  - UNICOR, Linhares, Espírito Santo
  - Hospital Anchieta, Brasília, Federal District
  - Hospital do Coração do Brasil, Brasília, Federal District
  - Hospital Felício Rocho, Belo Horizonte, Minas Gerais
  - Hospital Lifecenter, Belo Horizonte, Minas Gerais
  - Santa Casa de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Universidade Federal do Triangulo Mineiro, Uberaba, Minas Gerais
  - Instituto do Coração do Triângulo Mineiro, Uberlândia, Minas Gerais
  - Cardiocenter, João Pessoa, Paraíba
  - Centro Integrado de Medicina Intervencionista, Belém, Pará
  - Hospital Agamenon Magalhães, Recife, Pernambuco
  - Procape, Recife, Pernambuco
  - Fundação Universitária de Cardiologia, Porto Alegre, Rio Grande do Sul
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUC, Porto Alegre, Rio Grande do Sul
  - Santa Casa de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Santa Isabel, Blumenau, Santa Catarina
  - Instituto de Cardiologia de Santa Catarina, Florianópolis, Santa Catarina
  - Cardiologia Catanduva, Catanduva, São Paulo
  - Santa Casa de Limeira, Limeira, São Paulo
  - Santa Casa de Marília, Marília, São Paulo
  - INCORPI - Hosp. Fornecedores de Cana, Piracicaba, São Paulo
  - Santa Casa de São Carlos, São Carlos, São Paulo
  - Fundação Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - Hospital Bandeirantes, São Paulo, São Paulo
  - Hospital Beneficência Portuguesa, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo
  - Instituto de Assistencia Médica ao Sevidor Público Estadual- IAMSPE, São Paulo, São Paulo
  - EMCOR Emergências do Coração, Piracicaba, São Paulo - SP
  - Hospital das Clínicas de Ribeirão Preto, Ribeirão Preto, São Paulo - SP
  - INTERVECENTER Serviços Cardiovasculares, Palmas, Tocantins

REFERENCES:
- [Derived] Feres F, Costa RA, Abizaid A, Leon MB, Marin-Neto JA, Botelho RV, King SB 3rd, Negoita M, Liu M, de Paula JE, Mangione JA, Meireles GX, Castello HJ Jr, Nicolela EL Jr, Perin MA, Devito FS, Labrunie A, Salvadori D Jr, Gusmao M, Staico R, Costa JR Jr, de Castro JP, Abizaid AS, Bhatt DL; OPTIMIZE Trial Investigators. Three vs twelve months of dual antiplatelet therapy after zotarolimus-eluting stents: the OPTIMIZE randomized trial. JAMA. 2013 Dec 18;310(23):2510-22. doi: 10.1001/jama.2013.282183. PMID 24177257
- [Derived] Feres F, Costa RA, Bhatt DL, Leon MB, Botelho RV, King SB 3rd, de Paula JE, Mangione JA, Salvadori D Jr, Gusmao MO, Castello H Jr, Nicolela E Jr, Perin MA, Devito FS, Marin-Neto JA, Abizaid A. Optimized duration of clopidogrel therapy following treatment with the Endeavor zotarolimus-eluting stent in real-world clinical practice (OPTIMIZE) trial: rationale and design of a large-scale, randomized, multicenter study. Am Heart J. 2012 Dec;164(6):810-6.e3. doi: 10.1016/j.ahj.2012.09.009. Epub 2012 Nov 14. PMID 23194480